CLINICAL TRIAL: NCT02909361
Title: A Multicenter, Prospective, Real-world Study to Evaluate the Safety Profile and Effectiveness in Chinese Patients Who Received Fulvestrant 500mg as First-line Endocrine Treatment for Advanced Breast Cancer
Brief Title: Fulvestrant 500mg in Patients With Advanced Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xichun Hu, Director of department of medical oncology, Fudan University
Other Study IDs: Fudan BR2016-21
Record Dates: First submitted 2016-09-12; First posted 2016-09-21 (Estimated); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 53 Months
Biospecimen Retention: Samples With DNA — Plasma Sample will be collected at the time of study start and discontinuation base on the clinical practice.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Fulvestrant: 500 mg on days 0, 14, and 28, and every 28 days thereafter
  Interventions: Drug: Fulvestrant

INTERVENTIONS:
Drug: Fulvestrant — 500 mg on days 0, 14, and 28, and every 28 days thereafter
  Other Names: Fulvestrant Injection

SUMMARY:
Fulvestrant 500mg in Patients With Advanced Breast Cancer

DETAILED DESCRIPTION:
A multicenter, prospective study real-world to evaluate the safety profile and effectiveness in Chinese patients who received Fulvestrant 500mg as first-line endocrine treatment for Advanced breast cancer

ELIGIBILITY:
Inclusion Criteria:

1. Chinese women with estrogen receptor positive, locally advanced or metastatic breast cancer who has already received Fulvestant 500mg treatment as determined by treating physician. Ovarian suppression in premenopausal women is permitted, including ovarian ablation and LHRHa.
2. Histologically confirmed positive oestrogen receptor status (ER positive) of primary breast cancer or metastatic tumour tissue, according to the local laboratory parameters.
3. Prior endocrine therapy for advanced disease was not permitted.
4. The prescription of the Fulvestant is clearly separated from the decision to include the subject in the NIS, and is part of normal medical practice. The recruitment of the patient to the study should be within 1 month of the first Fulvestant injection.
5. Provision of subject informed consent.

Exclusion Criteria:

1. If participating in any controlled clinical trial, the subject cannot take part in this study.
2. HER2 overexpression or gene amplification, ie, immunohistochemistry (IHC) 3+ or fluorescence in situ hybridisation (FISH)+, where appropriate.
3. Pervious regimen of endocrine therapy for advanced disease.
4. More than one regimen of chemotherapy for advanced disease.
5. Pregnancy and lactation.
6. Severe hepatic impairment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese women with estrogen receptor positive, locally advanced or metastatic breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-10-11 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Incidence, nature and severity of all Adverse Events assessed by CTCAE V4.0 | From date of randomization until the date of date of death from any cause or last visit, assessed up to 100 months.
  Incidence, nature and severity of all Adverse Events assessed by CTCAE V4.0

SECONDARY OUTCOMES:
ORR | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.
  Objective Response Rate
CBR | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.
  Clinical Benefit Rate
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.
  Progression Free Survival
OS | From date of randomization until the date of date of death from any cause or last visit, assessed up to 100 months.
  Overall Survival

CONTACTS AND LOCATIONS:
Overall Officials: Xichun Hu, MD, PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, China